CLINICAL TRIAL: NCT06377371
Title: A Pilot Study to Evaluate Feasibility of Intraoperative Tracing of Meningioma Using [Cu64]DOTATATE
Brief Title: Feasibility of Intraoperative Tracing of Meningioma Using [Cu64]DOTATATE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Curium US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-03025815
Record Dates: First submitted 2024-04-10; First posted 2024-04-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with MRI findings compatible with meningioma who have an indication for surgery (Experimental): A diagnostic intervention in which patients will undergo intraoperative meningioma tracing using [Cu64]DOTATATE.
  Interventions: Diagnostic Test: Brain Imaging with [Cu64]DOTATATE; Procedure: Radio-guided Surgery With Neoprobe Utilization

INTERVENTIONS:
Diagnostic Test: Brain Imaging with [Cu64]DOTATATE — Patients will undergo a [Cu64]DOTATATE PET/MRI or PET/CT before undergoing radio- guided surgery. Patients will undergo another [Cu64]DOTATATE PET/MRI or PET/CT 6 weeks- 3 months after their surgery, and 6 months- 12 months after surgery.
Procedure: Radio-guided Surgery With Neoprobe Utilization — After the subjects undergo the preoperative [Cu64]DOTATATE PET/MRI, subjects will undergo radio-guided surgery in which the surgeon will utilize a standard intraoperative gamma probe (Neoprobe Gamma Detection System ®) to assess primary/residual tumor detection.

SUMMARY:
The study team hypothesizes that it is feasible to intraoperatively detect tumor following [CU64]DOTATATE injection using the gamma probe device.

DETAILED DESCRIPTION:
Objectives:

Primary objectives: The primary objective of this pilot study is to evaluate the feasibility of intraoperative tumor detection using [Cu64]DOTATATE. The study team further wants to validate the gamma count measurements using pre- and post-operative Positron Emission Tomography (PET) standardized uptake value (SUV) .

Secondary Objectives: To correlate intraoperative tracing findings with from pathology markers ( World Health Organization grade (WHO grade), Ki-67, Somatostatin Receptor 2 expression (SSTR2A expression), Estrogen receptor expression (ER expression), Progesterone receptor expression (PR expression)) using samples obtained as part of routine surgical care. To evaluate the correlation of post resection gamma count with longitudinal PET follow up.

Exploratory objectives: To establish best practices for integration of intraoperative tumor tracing using the neoprobe into the surgical workflow. To determine surgical candidates who will benefit most from intraoperative tracing based on tumor location, MRI features, etc.

Overall Design:

This is a single-center prospective observational pilot study to determine the feasibility of using [Cu64]DOTATATE for intraoperative tumor detection. 20 patients diagnosed with meningioma by conventional magnetic resonance imaging (MRI) who are candidates for surgical resection will be enrolled. Enrollment will be facilitated by colleagues in the neurosurgery department (also co- investigators on this study) with whom the PI has had several years of collaboration and an ongoing referral stream (6pprox.. 5 patients per week).

Patients will subsequently undergo pre-operative [Cu64]DOTATATE PET/MRI 12-24 hours prior to surgery. Given that [Cu64]DOTATATE has a much longer half-life compared to [Ga68]DOTATATE, it is uniquely suited for this application, allowing the patient to be injected once with the clinically approved dose, undergo immediate Positron Emission tomography scan and magnetic resonance imaging scan (PET/MRI) or Positron Emission tomography scan and computed tomography scan (PET/CT), and undergo resection the following day with sufficient radiotracer in situ for radio-guided surgery (RGS).

During the operation, the neurosurgeon will make a number of measurements using the neoprobe (available at our institution and currently in frequent routine clinical use for intraoperative sentinel node detection; commonly used for breast cancer, melanoma, oral cancer):

1. After exposing the tumor, and immediately before removal, tumor counts will be documented with the neoprobe. This count will be correlated with preoperative [Cu64]DOTATATE SUV to evaluate the relationship between radiographic radiotracer uptake and intraoperative radioactivity of the tumor.
2. After removing all tumor that can be removed safely, the surgeon will grade whether they feel they obtained a gross total resection (GTR) or whether tumor was left behind (subtotal resection (STR), e.g. because the surgeon had to leave behind tumor attached to critical structure). In case of STR, the neoprobe will be used to measure counts in the remaining tumor. In case of presumed GTR, the neoprobe will be used to measure counts in the resection cavity. This second count will be correlated with post-operative [Cu64]DOTATATE SUV to evaluate the effectiveness of this method in evaluating residual tumor.

These steps will not alter the regular course of the surgery in any way. Patients will have two follow-up points after the surgery: 1) at 6 weeks to 3 months post-op and 2) at 6 months to 12 months post-op. Patients will be clinically examined and will undergo repeat [Cu64]DOTATATE PET/MRI or PET/CT during these follow up visits, as standard of care, with radiotracer dosage being funded by the study for the 1st follow up scan, and determined standard of care for the 2nd follow up scan.

ELIGIBILITY:
Inclusion Criteria:

* High suspicion of meningioma necessitating surgical resection based on conventional MRI criteria, or diagnosis of meningioma based on pathology reports from prior resection with radiographic findings of suspected recurrent or residual tumor necessitating repeat surgery.

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients undergoing endoscopic endonasal resection, eyebrow incision surgery, or any surgical procedure in which the neoprobe cannot be employed
* Patients with hypersensitivity to somatostatin analogs
* Patients with contraindications to conventional MRI
* Patients with prior history of cranial radiation therapy
* Patients currently enrolled in other therapeutic clinical trials related to meningioma will be excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative [Cu64]DOTATATE PET SUV | At time of enrollment
  preoperative lesion [Cu64]DOTATATE PET SUV
1st Post-operative [Cu64]DOTATATE PET SUV | 3 months
  6 weeks to 3 months follow up post operative [Cu64]DOTATATE PET SUV
2nd Post-operative [Cu64]DOTATATE PET SUV | 1 year
  6 months to 12 months follow up post operative [Cu64]DOTATATE PET SUV
MRI Size Measurements | At time of enrollment
  preoperative size measurements based on Response Assessment in Neuro-Oncology (RANO) guidelines
GTR vs STR Assessment | 6 weeks- 3 months
  postoperative MRI-based assessment of GTR versus STR by a neuroradiologist, as determined by the presence or absence of nodular dural-based enhancement on post contrast 3D T1-weighted MR imaging and direct comparison to preoperative MRI.
MRI Progression Assessment | 6-12 months
  follow-up MRI assessment of progression based on RANO guidelines
Target Lesion Neoprobe Count | At time of enrollment
  Neoprobe count of the target lesion prior to resection.
Subtotal Neoprobe Count | At time of enrollment
  Neoprobe count of the subtotally resected tumor or the resection cavity in case of presumed GTR post resection.
Reference Background Neoprobe Count | At time of enrollment
  Neoprobe count of the reference background measured at least 1 cm away from the tumor (measured in at least two locations depending on the operative field)

SECONDARY OUTCOMES:
SSTR2 expression | At time of clinical neuropathological evaluation of resected tumor tissue (Immediate postoperative setting).
  immunohistochemistry analysis of SSTR2 expression in the resected tumor
WHO grade | At time of clinical neuropathological evaluation of resected tumor tissue (Immediate postoperative setting).
  determined histomorphologically based on pathologist's assessment of resected tumor tissue.
Ki67 Proliferation Index | At time of clinical neuropathological evaluation of resected tumor tissue (Immediate postoperative setting).
  Ki67 Proliferation Index (percentage of positively stained tumor cells among the total number of malignant cells assessed).
ER/PR expression | At time of clinical neuropathological evaluation of resected tumor tissue (Immediate postoperative setting).
  determined based on pathologist's assessment of resected tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Ivanidze, MD/PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York-Presbyterian/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No